CLINICAL TRIAL: NCT04772729
Title: Does the Use of Faster Insulin Aspart vs. Aspart Lead to the Prolonged Glycemic Time in Range in Children Suffering From Type 1 Diabetes Who Use Continuous Glucose Monitoring?
Brief Title: Does the Use of Fiasp vs. Asp Lead to the Prolonged TIR in Children With Type 1 Diabetes?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TIR: Fiasp vs. Asp
Record Dates: First submitted 2021-01-25; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Diabetes type1; Diabetes Mellitus, Type 1
Keywords: CGM; continuous glucose monitoring system; TIR; Time In Range; insulin aspart; insulin faster aspart
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: A cross-over, open-label, randomized study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Aspart (Active Comparator): Patients will use the continuous subcutaneous insulin infusion of insulin aspart (Novo Rapid, Novo Nordisk) and RT-CGM for 4 weeks.
  Interventions: Drug: Insulin faster aspart (Fiasp, Novo Nordisk)
- Insulin Fiasp (Experimental): Patients will use the continuous subcutaneous insulin infusion of insulin faster aspart (Fiasp, Novo Nordisk) and RT-CGM for 4 weeks.
  Interventions: Drug: Insulin faster aspart (Fiasp, Novo Nordisk)

INTERVENTIONS:
Drug: Insulin faster aspart (Fiasp, Novo Nordisk) — Duration of the study: 10 weeks.
  It is assumed that the patients will attend 4 visits in Pediatric Diabetology Clinic, and 3 telephone consultations.
  W0: The study will start with a 2-week run-in period in order to normalize glycemia.
  W1: RT-CGM will be inserted. Subsequently, the participants will be randomly assigned to one of two groups (Fa-A or A-Fa), basing on which the order of insulin use will be determined.
  W2: after 2 weeks, diabetology telephone consultation (washout period).
  W3: after 2 weeks, diabetology consultation. Changing insulin type according to the allocation.
  W4: after 2 weeks, diabetology telephone consultation (washout period).
  W5: after 2 weeks, diabetology telephone consultation.
  W6: the results obtained throughout the study will be discussed with the patient and the parent.
  Other Names: Insulin aspart (Novo Rapid, Novo Nordisk)

SUMMARY:
The aim of the study is to assess whether the implementation of faster insulin aspart in children with Type 1 diabetes treated with intensive insulin therapy with the use of an insulin pump and using Real Time Continuous Glucose Monitoring (RT-CGM) systems leads to prolonged time in range (TIR) compared to insulin aspart.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 year of a history of type 1 diabetes;
* treatment with intensive insulin therapy with the use of an insulin pump (continuous subcutaneous insulin infusion, CSII) ≥3 months;
* using continuous glucose monitoring system for at least 1 month;
* HbA1c<8%;
* consent to participate in the study obtained from the parent and the patient (>16 years of age).

Exclusion Criteria:

* diabetes treated with multiple insulin injections with insulin pens (Multiple Daily Injections, MDI);
* concomitant medical problems which might significantly affect glucose levels;
* the withdrawal of the consent to participate in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Glycaemia difference in time in range (TIR) 70-180mg/dl | at week 4 of the study
Glycaemia difference in time in range (TIR) 70-180mg/dl | at week 8 of the study

SECONDARY OUTCOMES:
Glycaemia difference in time below range (TBR) | at weeks 4 and 8 of the study
Glycaemia difference in time above range (TAR) | at weeks 4 and 8 of the study
Glycaemia difference in the coefficient of variation (CV) | at weeks 4 and 8 of the study
Difference in the average glycemia levels + standard deviation | at weeks 4 and 8 of the study
Difference in Total Daily Dose (TDD) of insulin | at weeks 4 and 8 of the study
Difference in the basal rate of insulin | at weeks 4 and 8 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, Prof., Study Chair — Department of Pediatric Diabetology and Pediatrics, Pediatric Teaching Clinical Hospital of the Medical University of Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No